CLINICAL TRIAL: NCT01094106
Title: Local Infiltration Analgesia for Postoperative Pain After Caesarean Section. A Prospective, Randomised, Controlled Trial
Brief Title: Infiltration Analgesia After Caesarean Section
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: North Karelia Central Hospital (Other)
Responsible Party: Principal Investigator, Sanna Kouhia, MD, North Karelia Central Hospital
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: NCCHAne001
Record Dates: First submitted 2010-03-12; First posted 2010-03-26 (Estimated); Results first posted 2020-08-18 (Actual); Last update posted 2020-08-18 (Actual); Status verified 2020-08

CONDITIONS: Pain, Postoperative; Caesarean Section
Keywords: postoperative pain; infiltration analgesia; ropivacaine; Caesarean Section
MeSH Terms: conditions — Pain, Postoperative

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Ropivacaine 0,75% (Active Comparator): Postoperative wound infusion 15 mg /h / 48h
  Interventions: Drug: Ropivacaine 0,75%
- NaCl 0,9% (Placebo Comparator): Postoperative wound infusion with NaCl 0,9% 2 ml /h /48h
  Interventions: Drug: NaCl 0,9%

INTERVENTIONS:
Drug: Ropivacaine 0,75% — Postoperative wound infusion 2 ml/ h/ 48h
  Arms: Ropivacaine 0,75%
Drug: NaCl 0,9% — Postoperative wound infusion 2 ml/h/48h
  Arms: NaCl 0,9%

SUMMARY:
Infiltration of a local anesthetic into the surgical wound is a simple method to strive to control postoperative pain after surgery. In the investigators institution, this method is used quite often. However, there is a controversy regarding the analgesic efficacy. Moreover, the cost of the single use elastomeric pump used with this procedure is clearly higher than the costs of other routinely used analgesic methods.

According to the investigators observations, infiltration of a local anesthetic into the surgical wound after caesarean section seems to reduce the need for rescue analgesics. However, the scientific evidence of the efficacy of this technique is weak. The investigators decided to conduct a prospective, controlled, randomised, double blind trial on this topic.

The hypothesis is that wound infiltration with local anesthetic will reduce postoperative pain and opioid consumption after caesarean section without major adverse effects.

ELIGIBILITY:
Inclusion Criteria:

* volunteer
* age over 18 years
* spinal anesthesia
* ASA 1-2
* no allergy to used medications
* no medications which have effect on pain perception

Exclusion Criteria:

* patient's refusal to participate
* marked systemic disease

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 70 (Actual)
Dates: Start 2010-04; Primary Completion 2011-10 (Actual); Study Completion 2011-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Sakari Syväoja, MD, Principal Investigator — North Carelia CH, Department of Anesthesia
Locations (1):
- North Karelia Central hospital, Joensuu, Finland

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Three patients were excluded after recruitment and randomisation, for the following reasons: For one patient, an emergency operation was needed before the scheduled operation time; for one patient, the hospital pharmacy was unable to provide the study drug in time, and for one patient, no study drug was initiated because of communication errors.
Period: Overall Study
Arm/Group | Ropivacaine 0,75% | NaCl 0,9%
Started | 33 | 34
Completed | 33 | 34
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Ropivacaine 0,75%: Patients undergoing caesarean section under spinal anaesthesia
  Ropivacaine 0,75%: Postoperative wound infusion; initial bolus of 10 ml, followed by an infusion of 2 ml/ h/ 48h
- NaCl 0,9%: Patients undergoing caesarean section under spinal anaesthesia
  NaCl 0,9%: Postoperative wound infusion; initial bolus of 10 ml, followed by an infusion of 2 ml/h/48h
- Total: Total of all reporting groups
Arm/Group | Ropivacaine 0,75% | NaCl 0,9% | Total
Number analyzed (Participants) | 33 | 34 | 67
Age, Continuous [Mean (Standard Deviation); unit: years] | 30.1 (5.7) | 30.9 (5.7) | 30.5 (5.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 33 | 34 | 67
  Male | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  Finland | 33 | 34 | 67
Weight, kg [Mean (Standard Deviation); unit: kg] | 75.8 (12.6) | 80.6 (17.2) | 78.2 (15.2)
Height, cm [Mean (Standard Deviation); unit: cm] | 162.4 (5.7) | 162.9 (6.4) | 162.6 (6.0)
Dose of spinal bupivacaine, mg [Mean (Standard Deviation); unit: mg] | 11.9 (0.8) | 11.7 (0.8) | 11.8 (0.8)
Length of operation, min [Mean (Standard Deviation); unit: min] | 50.6 (18.3) | 46.6 (13.8) | 47.0 (16.2)

OUTCOME MEASURES:

1. Primary Outcome: The Demand of Rescue Analgesics (Oxycodone)
Description: The amount of oxycodone required 48 hours after operation. Oxycodone was administered when the strength of pain is over 3 on numeric rating scale (NRS) 0-10.
Time Frame: 48 hours
Measure: Mean (Standard Deviation); unit: mg
Arm/Group | Ropivacaine 0,75% | NaCl 0,9%
Number analyzed (Participants) | 33 | 34
mg | 47.5 (20.9) | 57.8 (29.4)
Statistical Analysis 1: Comparison: Ropivacaine 0,75% vs NaCl 0,9%; In a previous non-randomised study at our institution, the mean oxycodone consumption in the control group was 60.7 mg (SD, 22.2 mg) during the first 48 h after caesarean section. At α = 0.05, 31 patients would be needed in each group to achieve a power of 90% for detecting a 30% reduction in the need for rescue opioids, which we considered a clinically meaningful effect. We decided to enrol 70 patients. The final study population was 67 patients; Test type: Superiority; p = 0.10, t-test, 2 sided

2. Secondary Outcome: Strength of Pain on Numerical Rating Scale (NRS)
Description: Intensity of pain was recorded on a numerical rating scale (0-10), where higher scores mean more severe pain, during rest and when moving, for five time intervals (0-6 h, 6-12 h, 12-24 h, 24-36 h and 36-48 h); for each time interval, the highest recorded pain score was taken into account.
Time Frame: 48 hours, divided to five time intervals (0-6 h, 6-12 h, 12-24 h, 24-36 h and 36-48 h)
Measure: Median (Inter-Quartile Range); unit: units on a scale
Arm/Group | Ropivacaine 0,75% | NaCl 0,9%
Number analyzed (Participants) | 33 | 34
units on a scale
  Highest recorded pain scores at rest, 0-6 h | 5 [3 to 6] | 6 [4 to 7]
  Highest recorded pain scores at rest, 6-12 h | 3 [2 to 5] | 3.75 [2 to 5]
  Highest recorded pain scores at rest, 12-24 h | 3 [2 to 4] | 3 [1.5 to 5]
  Highest recorded pain scores at rest, 24-36 h | 2.25 [1 to 5] | 3 [2 to 4]
  Highest recorded pain scores at rest, 36-48 h | 1 [0 to 2] | 2 [0 to 4]
  Highest recorded pain scores when moving, 0-6 h | 6.5 [5 to 8] | 7 [5 to 8]
  Highest recorded pain scores when moving, 6-12 h | 5 [4 to 7] | 6 [4 to 7]
  Highest recorded pain scores when moving, 12-24 h | 5 [4 to 7] | 5.75 [4 to 6.5]
  Highest recorded pain scores when moving, 24-36 h | 4.25 [3 to 6] | 5 [3 to 6]
  Highest recorded pain scores when moving, 36-48 h | 3 [2 to 4.5] | 4 [3 to 6]
Statistical Analysis 1: Comparison: Ropivacaine 0,75% vs NaCl 0,9%; Highest recorded pain scores at rest, 0-6 h; Test type: Superiority; p = 0.08, Wilcoxon (Mann-Whitney) — No adjustments for multiple comparisons
Statistical Analysis 2: Comparison: Ropivacaine 0,75% vs NaCl 0,9%; Highest recorded pain scores at rest, 6-12 h; Test type: Superiority; p = 0.86, Wilcoxon (Mann-Whitney) — No adjustments for multiple comparisons
Statistical Analysis 3: Comparison: Ropivacaine 0,75% vs NaCl 0,9%; Highest recorded pain scores at rest, 12-24 h; Test type: Superiority; p = 0.66, Wilcoxon (Mann-Whitney) — No adjustments for multiple comparisons
Statistical Analysis 4: Comparison: Ropivacaine 0,75% vs NaCl 0,9%; Highest recorded pain scores at rest, 24-36 h; Test type: Superiority; p = 0.79, Wilcoxon (Mann-Whitney) — No adjustments for multiple comparisons
Statistical Analysis 5: Comparison: Ropivacaine 0,75% vs NaCl 0,9%; Highest recorded pain scores at rest, 36-48 h; Test type: Superiority; p = 0.20, Wilcoxon (Mann-Whitney) — No adjustments for multiple comparisons
Statistical Analysis 6: Comparison: Ropivacaine 0,75% vs NaCl 0,9%; Highest recorded pain scores when moving, 0-6 h; Test type: Superiority; p = 0.36, Wilcoxon (Mann-Whitney) — No adjustments for multiple comparisons
Statistical Analysis 7: Comparison: Ropivacaine 0,75% vs NaCl 0,9%; Highest recorded pain scores when moving, 6-12 h; Test type: Superiority; p = 0.43, Wilcoxon (Mann-Whitney) — No adjustments for multiple comparisons
Statistical Analysis 8: Comparison: Ropivacaine 0,75% vs NaCl 0,9%; Highest recorded pain scores when moving, 12-24 h; Test type: Superiority; p = 0.68, Wilcoxon (Mann-Whitney) — No adjustments for multiple comparisons
Statistical Analysis 9: Comparison: Ropivacaine 0,75% vs NaCl 0,9%; Highest recorded pain scores when moving, 24-36 h; Test type: Superiority; p = 0.37, Wilcoxon (Mann-Whitney) — No adjustments for multiple comparisons
Statistical Analysis 10: Comparison: Ropivacaine 0,75% vs NaCl 0,9%; Highest recorded pain scores when moving, 36-48 h; Test type: Superiority; p = 0.06, Wilcoxon (Mann-Whitney) — No adjustments for multiple comparisons

3. Secondary Outcome: Postoperative Nausea and Vomiting (PONV)
Description: The numbers of patients with at least mild nausea at any time post-operatively.
Time Frame: 48 hours
Measure: Number; unit: participants
Arm/Group | Ropivacaine 0,75% | NaCl 0,9%
Number analyzed (Participants) | 33 | 34
participants | 7 | 11
Statistical Analysis 1: Comparison: Ropivacaine 0,75% vs NaCl 0,9%; Test type: Superiority; p = 0.30, Chi-squared

ADVERSE EVENTS:
Arm/Group | Ropivacaine 0,75% | NaCl 0,9%
Serious Adverse Events (participants affected / at risk) | 0/33 | 0/34
Other Adverse Events (participants affected / at risk) | 1/33 | 2/34
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Ropivacaine 0,75% (N=33) | NaCl 0,9% (N=34)
Wound dressings becoming unpleasantly wet, resulting in termination of the study drug infusion (Skin and subcutaneous tissue disorders) | 1 | 1
Smarting of the wound (Skin and subcutaneous tissue disorders) | 0 | 1 — Smarting of the wound, necessitating termination of the study drug infusion

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes